CLINICAL TRIAL: NCT05399537
Title: A Safety Evaluation of Prismocitrate 18 in Patients Receiving Continuous Renal Replacement Therapy (CRRT)
Brief Title: Safety Evaluation of Prismocitrate 18 in Patients Receiving CRRT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXU558476
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Regional Citrate Anticoagulation (RCA); Continuous Renal Replacement Therapy (CRRT); Acute Kidney Injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Prismocitrate 18 using the PrisMax System Version 3.x with calcium line accessory (Experimental): This is a single-arm study. Patients will receive regional citrate anticoagulation (RCA) with Prismocitrate 18 (investigational drug) during their CRRT treatment using the PrisMax System Version 3.x with calcium line accessory (investigational device).
  Interventions: Drug: Prismocitrate 18; Device: PrisMax System Version 3.x with calcium line accessory

INTERVENTIONS:
Drug: Prismocitrate 18 — Prismocitrate 18 solution (investigational drug) will be used in pre-dilution mode only; the rate of administration depends on the targeted citrate dose and the prescribed flow rate. The pre-filter infusion rate of Prismocitrate 18 solution will be indexed to the blood flow rate (BFR) to achieve a target blood citrate concentration of 3 mmol/L of blood. The flow rate for the anticoagulation of the extracorporeal circuit will be titrated to achieve a post-filter concentration of iCa of 0.25 to 0.35 mmol/L.
Device: PrisMax System Version 3.x with calcium line accessory — The RCA software on PrisMax System Version 3.x with calcium line accessory (investigational device) will be enabled to carefully guide the health practitioner for citrate dosing and calcium compensation.

SUMMARY:
Prismocitrate 18 is a continuous renal replacement therapy (CRRT) solution to be used as a renal replacement solution and as an anticoagulant to prevent blood clotting in the extracorporeal circuit. The delivery of CRRT therapy is provided by the PrisMax System which includes regional citrate anticoagulation (RCA) software to facilitate citrate and calcium compensation prescription.

The objectives of this study are: 1) to confirm the safety of Prismocitrate 18 in patients receiving CRRT using continuous venovenous hemodiafiltration (CVVHDF) or continuous venovenous hemofiltration (CVVH) and 2) to observe that the software and interface for the PrisMax System Version 3.x with calcium line accessory allows for implementation of regional citrate anticoagulation (RCA) (citrate and calcium dosing) during CRRT with Prismocitrate 18 and intended prescription.

The study period of the patient's CRRT will be up to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years of age
* Patients who are candidates for CRRT
* Patients expected to survive for at least 24 hours
* Patients with a contraindication to heparin or an increased risk of hemorrhage
* Patient and/or legally-authorized representative has signed a written informed consent form (ICF) per 21 CFR Part 50.55(e)

Exclusion Criteria:

* Patients with a known allergy to citrate or who have ever experienced an adverse reaction associated with citrate products, including patients with a prior history of citrate toxicity
* Patients with acute liver failure, defined by the occurrence of encephalopathy and hepatic synthetic dysfunction within 26 weeks of the first symptoms of liver disease and without evidence of chronic liver disease
* Patients with acute-on-chronic liver failure characterized by acute decompensation of cirrhosis and a Child-Pugh Liver Failure Score >10
* Patients with refractory shock and associated lactic acidosis (lactate >4 mmol/L)
* Patients with a systemic ionized calcium concentration outside the normal physiologic range (1.0 - 1.3 mmol/L), or outside of the laboratory reference range (Note: It is acceptable to provide calcium supplementation or treatment for hypercalcemia to achieve a normal physiologic range prior to therapy initiation)
* Female patients of childbearing potential who are pregnant or breastfeeding. (Note: All female patients, who have not undergone a hysterectomy, bilateral oophorectomy with or without hysterectomy, or has medically documented ovarian failure before study Screening must have a negative serum beta human chorionic gonadotropic [B-hCG] pregnancy test at Screening)
* Patients who are currently participating in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with symptomatic hypocalcemia related to Prismocitrate 18 administration | Day 1 up to Day 10
  Defined as symptomatic patients (e.g., tetany/spasms, seizures, or cardiac events secondary to a prolonged QT interval), with symptoms deemed attributable to hypocalcemia and with a confirmed systemic ionized calcium < 0.9 mmol/L.
Number of participants with symptomatic hypercalcemia related to Prismocitrate 18 administration | Day 1 up to Day 10
  Defined as symptomatic patients (e.g., changes in mental status not explained by the interventions or underlying conditions or cardiac events secondary to a shortened QT interval), with symptoms deemed attributable to hypercalcemia and with a confirmed systemic ionized calcium > 1.4 mmol/L.
Number of participants with symptomatic citrate accumulation related to Prismocitrate 18 administration | Day 1 up to Day 10
  Defined as symptomatic patients (e.g., refractory acidosis), with symptoms deemed attributable to citrate accumulation and with a systemic total calcium to ionized calcium ratio > 2.5.

SECONDARY OUTCOMES:
Number of participants with Adverse Events related to study product and/or procedure | Day 1 up to Day 28
  Incidence of AE and SAE's are also considered secondary outcome measures and will be reported in the Adverse Event section
Delivery of regional citrate anticoagulation (RCA) therapy using PrisMax System Version 3.x | Day 1 up to Day 10
  Percentage of complete RCA treatments according to protocol

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Alabama at Birmingham/UAB, Birmingham, Alabama
  - University of Southern California (USC) / Keck Hospital, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Bon Secours Mercy Health-Springfield Regional Medical Center, Springfield, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Lt. Col. Luke Weathers, Jr. VA Medical Center, Memphis, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - Gamma Medical Research, Inc / McAllen Medical Center, McAllen, Texas

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: The Sponsor is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, the Sponsor will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If the Sponsor agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of the Sponsor prior to the release of any data